CLINICAL TRIAL: NCT02692222
Title: Measurement of Pulse Pressure Variation (PPV) and Cardiac Output (CO) by a New Application for Android™ (Captesia™) : Comparison With PPV and CO Obtained by a Method of Transpulmonary Thermodilution.
Brief Title: Measurement of Pulse Pressure Variation and Cardiac Output by a New Application for Android™ (Captesia™)
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Céline Boudart, MD, Erasme University Hospital
Other Study IDs: B406201526827
Record Dates: First submitted 2016-02-10; First posted 2016-02-26 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Bypass
Keywords: pulse pressure variation monitoring; Captesia; cardiac output monitoring

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPV: This study will track changes in PPV and CO before and after of volume expansion, which goal is to change the cardiac output.
  Interventions: Other: Calculation of PPV and CO with two methods

INTERVENTIONS:
Other: Calculation of PPV and CO with two methods

SUMMARY:
This study test the agreement and accuracy of Pulse Pressure Variation (PPV) and Cardiac Output (CO) obtained by the Android application Capstesia™ against the gold standard : PPV and CO calculated by thermodilution.

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) remains a good predictor of fluid responsiveness in the OR. However, PPV can be time-consuming to calculate (manual determination), is not always displayed on monitoring screens nor reliable through visual assessment and needs additional devices to be displayed. A new Android application (Captesia) automatically calculates the PPV utilizing a digital photograph of the arterial waveform from the monitor. The application determines the PPV by selecting peaks and troughs of the arterial curve.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for coronary artery bypass

Exclusion Criteria:

* patients with arrhythmias like atrial fibrillation
* patients with valvular insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for coronary artery bypass
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
PPV | at time of surgery
  the Pulse Pressure Variation will be calculated by the Android Application (Captesia) and by the Picco before and after a meneuver of volume expansion, which goal is to change the cardiac output.

SECONDARY OUTCOMES:
CO | at time of surgery
  the Cardiac Output will be calculated by the Android Application (Captesia) and by thermodilution before and after of volume expansion, which goal is to change the cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Céline F Boudart, MD, Principal Investigator — Erasme Hospital Bruxelles; Alexandre Joosten, MD, Principal Investigator — Erasme Hospital Bruxelles
Locations (1):
- Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Background] Yang X, Du B. Does pulse pressure variation predict fluid responsiveness in critically ill patients? A systematic review and meta-analysis. Crit Care. 2014 Nov 27;18(6):650. doi: 10.1186/s13054-014-0650-6. PMID 25427970
- [Background] Cannesson M, Le Manach Y, Hofer CK, Goarin JP, Lehot JJ, Vallet B, Tavernier B. Assessing the diagnostic accuracy of pulse pressure variations for the prediction of fluid responsiveness: a "gray zone" approach. Anesthesiology. 2011 Aug;115(2):231-41. doi: 10.1097/ALN.0b013e318225b80a. PMID 21705869